CLINICAL TRIAL: NCT07007988
Title: An Open-Label, Multicenter Phase I Study to Evaluate the Safety, Efficacy, and Pharmacokinetic Characteristics of Intraperitoneal Perfusion With Docetaxel Polymeric Micelles for Injection in Patients With Malignant Ascites
Brief Title: A Phase I Study of SIM0388 in Participants With Malignant Ascites.
Acronym: SIM0388-101
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIM0388-101
Record Dates: First submitted 2025-05-16; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Malignant Ascites
Keywords: Malignant Ascites; Solid tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIM0388 Dose escalation-mono (Experimental): Sequential cohorts of increasing dose levels of SIM0388 will be evaluated as monotherapy
  Interventions: Drug: SIM0388
- SIM0388 Dose expansion (Experimental): Recommended Dose(s) of SIM0388 as determined from Dose escalation will be evaluated
  Interventions: Drug: SIM0388

INTERVENTIONS:
Drug: SIM0388 — Abdominal perfusion
  Arms: SIM0388 Dose escalation-mono
Drug: SIM0388 — Abdominal perfusion
  Arms: SIM0388 Dose expansion

SUMMARY:
Malignant Ascites is a common complication of malignant tumor. The objective of this study is to evaluate the safety, efficacy, and pharmacokinetic characteristics of intraperitoneal perfusion with Docetaxel Polymeric Micelles (SIM0388) for injection in patients with malignant ascites

DETAILED DESCRIPTION:
The study starts with a dose escalation part followed by a dose expansion part. The primary objective of the dose escalation part is to evaluate the safety and tolerability of SIM0388 peritoneal perfusion, and determine the Maximum tolerated dose (MTD) and/or the recommended dose(s) (RD) of SIM0388 peritoneal perfusion.

The primary objective of the dose expansion part is to evaluate the efficacy of SIM0388 intraperitoneal perfusion in the treatment of malignant ascites.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation and signature of informed consent form;.
* ≥ 18 years of age, male or female.
* Participants with histologically and/or cytologically confirmed advanced/metastatic solid tumors;.
* Failure of at least one line of standard systemic anti-tumor therapy, unsuitability for standard systemic therapy, or absence of standard systemic therapy options.
* Moderate or greater ascites confirmed by ultrasonography
* ECOG performance status of 0, 1or 2.
* Life expectancy ≥ 3 months.
* Adequate hematologic and organ function.
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test. WOCBP and male subjects agree to use adequate contraception.

Exclusion Criteria:

* Participant is currently participating or has participated in a study of an investigational agent or using an investigational device within 4 weeks of first dose of study treatment
* Prior history of intraperitoneal paclitaxel-based therapy.
* Use of strong CYP3A4 inhibitors or inducers within 7 days before the first dose or anticipated use during the study.
* Failure to recover from adverse events caused by prior interventions to ≤Grade 1
* Complete intestinal obstruction within 30 days prior to the first dose.
* Myocardial infarction within 6 months, current unstable angina, primary cardiomyopathy, cerebrovascular events, congestive heart failure, symptomatic coronary artery disease requiring medication, arrhythmia requiring medication, QTcF interval >470 ms, or uncontrolled hypertension.
* Uncontrolled primary brain tumors or CNS metastases.
* Active infection.
* Known history of HIV infection.
* Active hepatitis B or hepatitis C infection.
* Hypersensitivity to any active or inactive ingredient of SIM0388.
* Pregnant or lactating women.
* Any condition (medical history, disease, treatment, or lab abnormality) that may interfere with study results, impede full participation, or deemed by the investigator to contradict the subject's best interests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Dose escalation:Dose limited toxicity (DLT) | DLT observation period (up to 35 days)
  Dose-limiting toxicity(DLT)
Dose escalation phase: Adverse Events (AEs) and Serious Adverse Events (SAEs) | Through study completion, an average of 2 years
  Adverse events will be assessed by investigator(s) according to NCI-CTCAE v5.0.
Dose expansion phase：ORRa(Objective response rate in ascites) | Through study completion, an average of 2 years
  Ascites ORRa assessed according to WHO criteria
Dose expansion phase：TTPa (Time to progress in ascites) | Through study completion, an average of 2 years
  Ascites TTPa assessed according to WHO criteria
Dose expansion phase：PuFS (Puncture/drainage -free survival) | Through study completion, an average of 2 years
  PuFS

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Gobroad Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No